CLINICAL TRIAL: NCT07380451
Title: Modular Optimization of Psychotherapy for Individuals With Depression Complicated by Personality Dysfunction and Complex Trauma: A Pilot Study in the Chilean Public Health System
Brief Title: Modular Intervention for Depression Study
Acronym: MIND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: MIDAP Millennium Institute for Research in Depression and Personality (Unknown)
Responsible Party: Principal Investigator, Alex Behn, Associate Professor, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 240531010; 1251070 (Other Grant/Funding Number: ANID - FONDECYT)
Record Dates: First submitted 2025-12-29; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Major Depression
Keywords: Complicated Depression; Early Life Adversity; Personality Dysfunction
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group clinical trial in which eligible participants are assigned in a 1:1 ratio to either an algorithm-based personalized modular psychotherapy or usual individual psychotherapy. Participants receive only the intervention to which they are assigned, and outcomes are compared between groups over the course of treatment and follow-up.
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study uses blinded outcome assessment and blinded statistical analysis. Primary outcome assessors are masked to participants' treatment assignment. In addition, the statistical analyst is masked to treatment allocation and does not have access to treatment assignment information during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modular Psychotherapy (MIND) (Experimental): Participants assigned to the MIND arm receive a personalized modular psychotherapy designed for depression complicated by personality dysfunction and/or complex trauma. All participants receive a core evidence-based depression treatment, including behavioral activation, cognitive, and interpersonal psychotherapy strategies. Additional short therapy modules are selected and added based on each participant's baseline emotional and interpersonal functioning profile following a module assignment algorithm. These modules target specific areas: emotion regulation difficulties, sensitivity to rejection and interpersonal threat, social functioning problems. Treatment is delivered as weekly individual psychotherapy sessions, with the number and combination of modules tailored to individual clinical needs.
  Interventions: Behavioral: Modular Intervention for Depression Therapy (MIND Therapy)
- Treatment as Usual (TAU) (Active Comparator): Participants assigned to the treatment as usual (TAU) arm receive individual psychotherapy as typically provided in public community mental health centers in Chile. This treatment reflects routine clinical practice and may vary in therapeutic approach according to the therapist's usual orientation. Sessions are delivered individually and on a weekly basis, without the use of the modular psychotherapy protocol.
  Interventions: Behavioral: Psychotherapy as Usual (TAU)

INTERVENTIONS:
Behavioral: Modular Intervention for Depression Therapy (MIND Therapy) — The MIND intervention is an algorithm-based, personalized, modular psychotherapy for adults with depression complicated by personality dysfunction and/or complex trauma. All participants receive a core evidence-based depression treatment that includes behavioral activation, cognitive, and interpersonal psychotherapy strategies. Additional short therapy modules are selected based on each participant's baseline emotional, interpersonal, and self-related functioning profile, using a predefined clinical algorithm. These modules target specific difficulties such as emotion regulation problems (DBT Module), sensitivity to rejection and interpersonal threat (MBT and CBASP Modules), social functioning difficulties (Social Thinning Module). The type and number of modules are tailored to individual needs following an algorithm based on baseline measures (DERS, A-RSQ, OQ-45-IR). Treatment is delivered as weekly individual psychotherapy sessions.
  Other Names: Psychotherapy
  Arms: Modular Psychotherapy (MIND)
Behavioral: Psychotherapy as Usual (TAU) — Psychotherapy as usual (TAU) consists of individual psychotherapy delivered in public community mental health centers according to routine clinical practice. Treatment is provided weekly by trained clinicians and may vary in therapeutic orientation, techniques, and structure depending on the therapist and center. TAU is not guided by the modular psychotherapy protocol or algorithm used in the experimental intervention and reflects standard care available in the Chilean public mental health system.
  Other Names: Psychotherapy
  Arms: Treatment as Usual (TAU)

SUMMARY:
The goal of this psychotherapy clinical trial is to evaluate whether a algorithm-based personalized modular psychotherapy is more effective than usual individual psychotherapy in treating major depressive disorder complicated by personality dysfunction and/or complex trauma in adults aged 18 to 65 receiving care in the Chilean public mental health system.

The main questions it aims to answer are:

* Does algorithm-based modular psychotherapy lead to greater clinically significant reduction and remission of depressive symptoms compared to usual psychotherapy?
* Does algorithm-based modular psychotherapy lead to greater improvement in emotional regulation, interpersonal functioning, and self-related functioning, including changes observed in daily life?

Researchers will compare algorithm-based modular psychotherapy to usual individual psychotherapy provided in public community mental health centers to see if the modular, personalized approach results in better clinical outcomes, stronger therapeutic alliance, and higher treatment satisfaction.

Participants will:

* Be randomly assigned to receive either algorithm-based modular psychotherapy or usual individual psychotherapy
* Attend weekly individual psychotherapy sessions
* Complete structured diagnostic interviews and self-report questionnaires before, during, and after treatment
* Provide brief daily reports on mood, emotions, and interpersonal experiences using a smartphone before and after treatment

DETAILED DESCRIPTION:
This randomized controlled clinical trial evaluates an algorithm-based personalized modular psychotherapy designed for adults with major depressive disorder whose condition is complicated by long-standing emotional, interpersonal, and self-related difficulties associated with early life adversity or personality functioning problems. These individuals often have poorer outcomes with standard psychotherapeutic approaches offered in public mental health services.

The experimental intervention consists of a modular psychotherapy approach. All participants in this group receive a core, evidence-based depression treatment. Additional short therapy modules are added based on each participant's baseline clinical profile following a module-assignment algorithm, targeting specific difficulties such as problems with emotion regulation, sensitivity to rejection and interpersonal threat, difficulties in social functioning, or disturbances in self-concept and self-worth. The number and type of modules are personalized for each participant, allowing the treatment to be tailored while remaining feasible within routine public mental health care.

The comparison group receives usual individual psychotherapy, which reflects standard care provided in community mental health centers in Chile. These treatments are delivered weekly by trained clinicians and are not guided by the modular protocol.

150 adults aged 18 to 65 will be recruited from public mental health centers. Eligible participants have major depressive disorder along with evidence of personality-related dysfunction and/or moderate to severe early life trauma. Participants are randomly assigned in a 1:1 ratio to either modular psychotherapy or usual care.

The primary outcomes of the study are clinically meaningful reduction in depressive symptoms and remission from depression following treatment. Secondary outcomes include changes in emotional regulation, interpersonal functioning, daily emotional and interpersonal experiences assessed through brief smartphone-based daily reports, quality of the therapeutic alliance, and satisfaction with treatment from both patients and therapists.

The purpose of this pilot trial is to determine whether a personalized algorithm-based modular psychotherapy approach improves clinical and functional outcomes compared to usual psychotherapy for people with complex depression in the Chilean public health system, and to inform future implementation and scaling of personalized mental health interventions.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of major depressive disorder, defined as:

  * Positive diagnosis on the MINI diagnostic interview, and
  * PHQ-9 score greater than 10
* Evidence of personality dysfunction, defined as a score above the cutoff on the Level of Personality Functioning Scale-Brief Form (LPFS-BF 2.0).
* History of moderate to severe early life adversity, defined as elevated scores on at least one scale of the Childhood Trauma Questionnaire (CTQ), and/or clinically significant alterations in self-organization.
* Presence of at least one elevated domain of alteration of self-organization, including emotion regulation difficulties, interpersonal sensitivity, and/or interpersonal functioning problems, as assessed by standardized self-report measures (DERS, A-RSQ, OQ-45-IR).
* Receiving care at a participating public community mental health center in Chile.
* Ownership of a smartphone (Android or iOS) with internet access and an active data plan.
* Ability to provide written informed consent.

Exclusion Criteria:

* Acute suicide risk requiring immediate intensive intervention, as assessed by the MINI.
* Any severe psychiatric disorder other than major depressive disorder that is the primary clinical diagnosis, including:

  * Schizophrenia or other psychotic disorders
  * Bipolar I disorder
* Severe substance use disorder, active within the past 6 months.
* Diagnosis of post-traumatic stress disorder (PTSD) meeting full diagnostic criteria, as assessed by standardized instruments (ITEM and ITQ).
* Meeting diagnostic criteria for:

  * Antisocial personality disorder (two or more criteria), or
  * Borderline personality disorder with more than three diagnostic criteria
* Severe medical, cognitive, or psychosocial condition that would interfere with participation in weekly psychotherapy.
* Concurrent participation in another active psychotherapy or initiation/change of psychotropic medication during the study period, except for:

  * Stable antidepressant treatment
  * Medications prescribed for sleep
  * Benzodiazepines used only on an as-needed (PRN) basis.
* Inability to comply with study procedures or assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Depression remission. | Baseline (pre-intervention), end of treatment (session 15; approximately 3 months), and 3-month post-treatment (approximately 6 months after baseline assessment).
  Primary depression outcomes will be assessed using the MINI International Neuropsychiatric Interview. The MINI is a structured interview. Remission is defined as a negative MINI assessment for major depressive disorder.
Clinically significant symptom reduction | Baseline (pre-intervention), end of treatment (session 15; approximately 3 months), and 3-month post-treatment (approximately 6 months after baseline assessment).
  Clinically significant symptom reduction will be assessed using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 has a range between 0 and 27. Higher scores indicate more symptom severity. Clinically significant symptom reduction is defined as a reduction of at least 5 points on the PHQ-9 from baseline and a post-treatment PHQ-9 score ≤9.

SECONDARY OUTCOMES:
Emotional regulation difficulties | Baseline (pre-intervention); during treatment at sessions 5, 10, and 15; and 3-month post-treatment follow-up (approximately 6 months after baseline).
  Emotional regulation will be assessed using the Difficulties in Emotion Regulation Scale (DERS-E). The DERS has a range of 25 to 125. Higher scores indicate more emotion regulation difficulties.
Interpersonal sensitivity and rejection sensitivity | Baseline (pre-intervention); during treatment at sessions 5, 10, and 15; and 3-month post-treatment follow-up (approximately 6 months after baseline).
  Interpersonal sensitivity will be assessed using the Adult Rejection Sensitivity Questionnaire (A-RSQ). Changes in sensitivity to interpersonal rejection will be evaluated from baseline to post-treatment. The A-RSQ has a range of 1 to 36. Higher scores indicate more rejection sensitivity.
Interpersonal functioning and social problems | Baseline (pre-intervention); during treatment at sessions 5, 10, and 15; and 3-month post-treatment follow-up (approximately 6 months after baseline).
  Interpersonal functioning will be measured using the Interpersonal Relations subscale of the Outcome Questionnaire - Interpersonal Relations (OQ-45-IR). Changes in social and interpersonal problems will be assessed from baseline to post-treatment. The range of the OQ-45 is 0 to 44. Higher scores indicate more interpersonal problems.
Daily emotional and interpersonal functioning | One week prior to treatment initiation and one week following treatment completion (after 15 sessions; approximately 3 months after baseline assessment).
  Daily emotional and interpersonal functioning will be assessed using smartphone-based ecological momentary assessment (EMA). Participants will report momentary negative affect, interpersonal experiences, rejection sensitivity, and self-related experiences multiple times per day during one week before treatment and one week after treatment.
Therapeutic alliance | After each treatment session, from session 1 through session 15 (approximately 3 months)
  Therapeutic alliance will be assessed using the Working Alliance Inventory (WAI), completed by participants after each therapy session. Change in alliance quality over the course of treatment will be examined.The range of the WAI is 12 to 84. Higher scores indicate a better working alliance perceived by the patient.
Treatment satisfaction | End of treatment (after session 15; approximately 3 months after baseline)
  Treatment satisfaction will be assessed in patients using the Client Satisfaction Questionnaire-8 (CSQ-8). The range of the CSQ-8 is 8 to 32. Higher scores indicate more satisfaction with the treatment.
Improvements in Quality of life | Baseline (pre-intervention); during treatment at sessions 5, 10, and 15; and 3-month post-treatment follow-up (approximately 6 months after baseline).
  Quality of life will be assessed using the Recovering Quality of Life questionnaire (ReQoL). Changes in quality of life will be evaluated from baseline to post-treatment and follow-up. The range of the ReQoL is 0 to 40. Higher scores indicate better perceived quality of life.
Acceptability of the Intervention | End of treatment (after session 15; approximately 3 months after baseline)
  Therapist perspectives on the intervention will be assessed using the Acceptability of Intervention Measure (AIM). The range of the AIM is 0 to 5. Higher scores indicate more acceptability of the intervention.
Feasibility of Intervention | End of treatment (after session 15; approximately 3 months after baseline)
  Therapist perspectives on the feasibility of the intervention will be asses using the Feasibility of Intervention Measure (FIM). The range of the FIM is 0 to 5. Higher scores indicate that the intervention is considered more feasible by the therapists.
Intervention Appropriateness | End of treatment (after session 15; approximately 3 months after baseline)
  Therapist perspectives on the appropriateness of the intervention will be measured using the Intervention Appropriateness Measure (IAM). The range of the IAM is 0 to 5. Higher scores indicate higher intervention appropriateness.
Disability/Functional Impairment | Baseline (pre-intervention); during treatment at sessions 5, 10, and 15; and 3-month post-treatment follow-up (approximately 6 months after baseline).
  Patient's degree of disability and functional impairment will be assessed through the WHO Disability Assessment Schedule (WHODAS). The range of the WHODAS is 12 to 60. Higher scored indicates higher disability.
Personality Functioning | Baseline (pre-intervention); during treatment at sessions 5, 10, and 15; and 3-month post-treatment follow-up (approximately 6 months after baseline).
  Patient's personality functioning will be assess using the Levels of Personality Functioning Scale (LPFS-BF). The range of the LPFS is 12 to 48. Higher socres indicate more personality dysfunction.
Psychological Distress | Baseline (pre-intervention); during treatment at sessions 5, 10, and 15; and 3-month post-treatment follow-up (approximately 6 months after baseline).
  Patient's psychological distress will be assessed using the Clinical Outcomes in Routine Evaluation - Outcome Measure Short Version (CORE-10). The rage of the CORE-10 is 0,8 to 3,2. Higher scores indicate more psychological distress.

OTHER OUTCOMES:
Mentalizing Capacity | Baseline (pre-intervention); during treatment at sessions 5, 10, and 15; and 3-month post-treatment follow-up
  Patient's mentalizing capacity will be assess throughout the study using the Multidimensional Mentalizing Questionnaire (MMQ). The range of the MMQ is 1 to 5. Higher scores indicate higher mentalizing capacity.

CONTACTS AND LOCATIONS:
Locations (5):
- Chile (5):
  - CDT CASR, Santiago
  - COSAM La Bandera, Santiago
  - COSAM La Granja, Santiago
  - COSAM La Pintana, Santiago
  - COSAM Rinconada, Santiago

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared.